CLINICAL TRIAL: NCT06453941
Title: The Validation and Beneficial Effects of Yizhi Baduanjin for Patients With Mild Cognitive Impairment: a Pilot Randomised Controlled Trial
Brief Title: Yizhi Baduanjin for Patients With Cognitive Impairment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only 1 subject has been recruited.
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW23-082
Record Dates: First submitted 2023-04-10; First posted 2024-06-12 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Mild Cognitive Impairment (MCI); Alzheimers Disease (AD); Non-drug intervention; Baduanjin
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yizhi Baduanjin group (Experimental): The Yizhi Baduanjin group will practice Yizhi Baduanjin as intervention for 6 months, and the participants will be examined for assessment indicators on the 1st, 3rd, 6th month after the intervention started.
  Interventions: Other: Yizhi Baduanjin (Eight Pieces of Brocades for Mental Health Promotion)
- Control group (No Intervention): The control group has no intervention until 6 months after the intervention of the experimental group started, but the participants will be examined for the same assessment indicators together with the experimental group.

INTERVENTIONS:
Other: Yizhi Baduanjin (Eight Pieces of Brocades for Mental Health Promotion) — Yizhi Baduanjin (Eight Pieces of Brocades for Mental Health Promotion) is a newly compiled routine developed on the foundation of the traditional Baduanjin (Eight Pieces of Brocades), which is a traditional Chinese medical health exercise consisted of eight movements to be practiced by oneself.
  Arms: Yizhi Baduanjin group

SUMMARY:
The trial is designed to examine whether Yizhi Baduanjin could slow down and improve in memory, logical thinking and cerebral function in patients with mild cognitive impairment (MCI). 30 MCI patients will be recruited and randomly assigned to Yizhi Baduanjin intervention group control group for 6 months. The primary outcome is changes in Montreal Cognitive Assessment (MoCA) questionnaire; other outcome includes Cognitive Function Assessment questionnaire.

DETAILED DESCRIPTION:
Alzehimer Disease (AD), generally known as dementia, is system of pathological changes of the central nervous system, with the major symptoms of progressive memory loss, cognitive disorder, personality changes and difficulty speaking. Mild Cognitive Impairment (MCI) is always regarded as "prodromal AD", and as a stage of AD in the revised diagnostic guidelines. It is a condition with minor memory decline, and minor difficulties with attention and learning. MCI patients have a much higher risk of progress to AD than the general population. AD increases along with aging, while aging is a worsening global issue. The onset of AD is difficult to recognize, and the progression is non-reversible and without cure, while the intervention during the MCI stage would be effective for preventing the progression to AD. The pathogenesis of MCI is yet to be investigated, so the pharmaceuticals are under debate. The non-drug therapies have few side effects and are more acceptable to patients, The investigators believe that Yizhi Baduajin, a newly complied routine based on the traditional Chinese medical health practice Baduanjin, is a possible intervention to prevent MCI and AD which could be practiced for long-term. Therefore, this pilot controlled trial is proposed to verify the effect of Yizhi Baduanjin and investigate how it improve and promotes mental and cerebral functions, and to explore and develop a replicable model of Yizhi Baduanjin MCI service package that includes MCI screening and education, as well as the Yizhi Baduanjin teaching.

The hypothesis is that the progression of MCI patients who practice Yizhi Baduanjin will slow down and improve in memory, logical thinking and cerebral function than MCI patients who do not practice. Also, Yizhi Baduanjin is a more acceptable intervention for middle-aged and elderly people, it is also easier to popularize in replicable model at a lower cost.

The trial will recruit 30 participants, and divide randomly into two groups with 15 participants each. The experimental group will practice Yizhi Baduanjin as an intervention for 6 months, and the participants will be examined for assessment indicators on the 1st, 3rd, 6th month after the intervention starts. The control group has no intervention until 6 months after the intervention of the experimental group started, but the participants will be examined for the same assessment indicators together with the experimental group. The Montreal Cognitive Assessment (MoCA) questionnaire and Cognitive Function Assessment questionnaire will be used as the assessment instruments, and data collected from the two groups will be compared and assessed.

ELIGIBILITY:
Inclusion Criteria:

1. 60 to 75 years old.
2. Voluntarily and sign the informed consent form.
3. Non-handicapped, able to complete the cognitive function examination.
4. Fulfill the diagnostic criteria.
5. Montreal Cognitive Assessment (MoCA )Scale < 26

Exclusion Criteria:

1. Fail to meet the inclusion criteria.
2. Fail to comply to the requirements, or fail to complete the examination.
3. Unwilling or unable to learn and practice the Yizhi Baduanjin routine.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Changes in Montreal Cognitive Assessment (MoCA ) | Baseline, 1-month, 3-month, 6-month
  Questionnaire with 8 categories, 33 items with a total score of 30.

SECONDARY OUTCOMES:
Changes in Cognitive Function Assessment | Baseline, 1-month, 3-month, 6-month
  Questionnaire with 4 Categories, total items and scores vary according to participants' response.

CONTACTS AND LOCATIONS:
Overall Officials: Zhangjin Zhang, MMed, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No